CLINICAL TRIAL: NCT00270881
Title: Phase 1/2 Study of Cord Blood Transplantation From Unrelated Donor for Adult Patients With Hematologic Malignancies Using Myeloablative Conditioning Regimen
Brief Title: Safety and Efficacy of Unrelated Cord Blood Transplantation for Adult Patients With Hematologic Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Keio University (Other)
Responsible Party: Principal Investigator, Takehiko Mori, M.D., Ph.D., Dr., Keio University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSGCT-CB2005
Record Dates: First submitted 2005-12-28; First posted 2005-12-29 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Acute Myelogenous Leukemia; Acute Lymphoblastic Leukemia; Chronic Myelogenous Leukemia; Myelodysplastic Syndrome
Keywords: cord blood transplantation; myeloablative regimen; hematologic malignancies
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Hematologic Neoplasms | interventions — Cord Blood Stem Cell Transplantation; Cyclophosphamide; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Cord blood transplantation — unrelated cord blood transplantation
Radiation: TBI — Total body irradiation (TBI) 12Gy
Drug: cyclophosphamide — cyclophosphamide 120mg/kg
Drug: cytarabine — cytarabine 3g/m2x4

SUMMARY:
The primary purpose of this study is to evaluate the safety and efficacy of cord blood transplantation for adult patients with hematologic malignancies including refractory acute leukemia. The transplant procedure was determined in detail according to the previously published report showing a high survival, so that the investigators could expect a similar result.

DETAILED DESCRIPTION:
Although cord blood is considered as an alternative donor source for allogeneic hematopoietic stem cell transplantation, its procedure has yet to be standardized. Recently, a single institute result of cord blood transplantation for adult patients with hematologic malignancies have been reported by Takahashi et al (Blood 2004:104;3813-3820), in which the survival was significantly better than that of bone marrow transplantation from unrelated donor. The purpose of this study was to reevaluate the safety and efficacy of cord blood transplantation for adult patients with hematologic malignancies using the same transplant procedures in a multi-institutional setting.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute leukemia, chronic myelogenous leukemia, and myelodysplastic syndrome
* Lack of HLA-identical or 1 locus mismatched related donor
* Age over 20, and under 55
* Performance status 0 or 1
* No moderate or sever organ dysfunction (liver, kidney, heart, lungs)
* No anti-HLA antibody
* Informed consent was obtained

Exclusion Criteria:

* Uncontrollable diabetes
* Uncontrollable hypertension
* Active infection
* TPHA, HBs-Ag, HCV-Ab positive
* HTLV-I, HIV positive

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Non-relapse mortality at 1 year | 1 year

SECONDARY OUTCOMES:
Engraftment | day 56
Disease free survival | 1 year
Overall survival | 1 year
Incidence of acute and chronic graft-versus-host disease | day100 and 1 year
Incidence of infectious complication | 1year
Duration of hospitalization | 1 year
Immune reconstitution after transplantation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hisashi Sakamaki, M.D., Ph.D., Study Chair — Tokyo Metropolitan Komagome Hospital
Locations (1):
- Keio University School of Medicine, Tokyo, Japan